CLINICAL TRIAL: NCT07372625
Title: A Phase 1, Open-label, 2-part, Drug-Drug Interaction Study to Evaluate the Effects of Multiple Oral Doses of Rezatapopt on the Pharmacokinetics of Metformin, Rosuvastatin, Repaglinide, and Midazolam in Patients With Advanced Solid Tumors Harboring a TP53 Y220C Mutation.
Brief Title: A Study to Investigate the Effects of Multiple Doses of Rezatapopt on the Pharmacokinetics of Metformin, Rosuvastatin, Repaglinide, and Midazolam in Patients With Advanced Solid Tumors Harboring a TP53 Y220C Mutation.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PMV Pharmaceuticals, Inc (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PMV-586-106
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: TP53 Y220C Mutation; Advanced Solid Tumors
Keywords: Y220C; PC14586; PMV Pharma; PMV; rezatapopt; Phase 1; metformin; rosuvastatin; repaglinide; midazolam; DDI
MeSH Terms: interventions — Metformin; Tablets; Rosuvastatin Calcium; repaglinide

STUDY DESIGN:
Intervention Model Description: Each patient will serve as their own control for assessing the effects of multiple oral doses of rezatapopt on the PK of metformin, rosuvastatin, repaglinide, and midazolam. The study will comprise 2 parts: Part A (24-day DDI portion) will use a fixed-sequence design, comprising a screening period and 2 treatment periods and Part B (Cycle 1 through Cycle 33, rezatapopt only), which will administer rezatapopt in 21-day treatment cycles. In Part A Treatment Period 1, the PK of metformin, rosuvastatin, repaglinide, and midazolam will be evaluated when administered without rezatapopt. In Part A Treatment Period 2, the effects of rezatapopt on the PK of metformin, rosuvastatin, repaglinide, and midazolam will be evaluated. The PK of rezatapopt and its metabolites will also be assessed. Patients who complete Part A without suspected disease progression, unacceptable toxicity or another discontinuation criterion may continue to Part B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A, Days 1-24 and Part B, Cycles 1-33 (Experimental): Patients will receive a cocktail of metformin and rosuvastatin after a morning meal on Day 1. Serial PK samples will be collected on Days 1-3. Days 2-5 will serv as a washout period.
  On Day 2, patients will receive a cocktail of repaglinide and midazolam. Serial PK samples will be collected on Days 2-3. Days 3-5 will serve as a washout period.
  On Days 6-21 patients will receive rezatapopt with serial PK samples taken on Days 6-7 and sparse PK on Day 14.
  On Day 22, patients will receive rezatapopt concurrently with a cocktail of metformin and rosuvastatin. Serial PK samples will be collected on Days 22-24.
  On Day 23, patients will receive rezatapopt concurrently with a cocktail of repaglinide and midazolam. Serial PK samples will be collected on Days 23-24.
  In Part B, patients will receive rezatapopt as 2000 mg PO QD in 21-day cycles through Cycle 33 (approximately 2 years) or until another discontinuation criterion is met.
  Interventions: Drug: metformin hydrochloride 500 mg tablet; Drug: rosuvastatin 10 mg tablet; Drug: repaglinide 0.5 mg tablet; Drug: midazolam hydrochloride syrup; Drug: rezatapopt

INTERVENTIONS:
Drug: metformin hydrochloride 500 mg tablet — 500-mg immediate release tablet PO
Drug: rosuvastatin 10 mg tablet — 10-mg tablet PO
Drug: repaglinide 0.5 mg tablet — 0.5-mg tablet PO
Drug: midazolam hydrochloride syrup — 2 mg dose (5-mg/2.5 mL syrup) PO
Drug: rezatapopt — 2000 mg dose (4 x 500-mg tablets) PO

SUMMARY:
This study aims to evaluate the effects of rezatapopt on the pharmacokinetics of metformin, rosuvastatin, repaglinide, and midazolam in patients with advanced solid tumors harboring a TP53 Y220C mutation.

DETAILED DESCRIPTION:
Rezatapopt (PC14586) is a first-in-class oral, small molecule p53 reactivator that is selective for the TP53 Y220C mutation.

This Phase 1, open-label, drug-drug interaction study will investigate the effect of multiple oral doses of rezatapopt on the pharmacokinetics (PK) of metformin, rosuvastatin, repaglinide, and midazolam in patients with advanced solid tumors harboring a TP53 Y220C mutation. This study will consist of 2 parts, Part A and Part B.

Part A is a 24-day drug-drug interaction (DDI) portion that follows a fixed- sequence design, including a screening period and 2 treatment periods.

In Treatment Period 1 patients will receive metformin and rosuvastatin, followed by repaglinide and midazolam. Patients will not receive rezatapopt during Treatment Period 1.

Following washout, in Treatment Period 2 which will begin on Day 6, patients will receive 2000 mg rezatapopt administered orally once daily along with metformin and rosuvastatin, and then repaglinide and midazolam in accordance with the fixed-sequence dosing schedule. Serial PK samples will be collected on designated days throughout Part A.

Patients who complete Part A without suspected disease progression and unacceptable toxicity or another discontinuation criterion and who are deemed likely to continue benefiting from the study treatment, will be allowed to continue treatment with rezatapopt in Part B.

In Part B, patients will receive 2000 mg rezatapopt orally daily in 21-day cycles, up to Cycle 33 (approximately 2 years of rezatapopt treatment, inclusive of Part A) or until another discontinuation criterion is met.

A maximum of approximately 14 patients are planned to enroll in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. 18 years and older
3. ECOG performance status (PS) score of 0 or 1
4. Confirmed locally advanced or metastatic solid malignancy with a TP53 Y220C mutation identified through a tumor-tissue based (e.g., FoundationOneCDx, PathGroup, Caris WES, MSK IMPACT, TEMPUS) or a liquid-biopsy based (e.g., Caris, MSK Access) NGS molecular test.

   - Patients with primary CNS tumors are allowed to enroll
5. Patients with castration-resistant prostate cancer must have ongoing androgen deprivation therapy with a gonadotropin-releasing hormone analog or inhibitor or orchiectomy (medical or surgical castration)
6. Adequate organ function
7. Life expectancy ≥3 months as assessed by the Investigator

Exclusion Criteria:

1. Patients with ovarian, breast, lung, or endometrial tumors who are eligible for the PYNNACLE Phase 2 trial (NCT04585750), unless the corresponding cohort in the PYNNACLE trial is closed to enrollment at the time of screening (to avoid overlap with that study).
2. Treatment, food, or drink with any of the following:

   * Any systemic anticancer therapies, including but not limited to chemotherapy, small molecule, biologic, or hormonal agents from a previous treatment regimen, or investigational anticancer agents from clinical study within 21 days or 5 half-lives (whichever is longer) prior to the first dose of study drugs
   * Radiotherapy within 14 days of first dose of study drugs. Palliative radiotherapy particularly limited field and stereotactic body radiation therapy to non-target lesions should be allowed.
   * Inhibitors or inducers of the enzymes and transporters being tested in this study within 14 days of starting study drugs
   * Sensitive substrates of CYP3A4 or CYP2C8 with a narrow therapeutic index within 14 days of starting study drugs
   * Herbal preparations/medications known to be strong or moderate CYP3A4 inhibitors or inducers or to have other significant potential for interaction with rezatapopt within 14 days of starting study drugs
   * Foods or drinks with CYP3A inhibition potential (e.g., grapefruit, grapefruit juice, Seville orange juice, pomelos, starfruits) within 14 days of starting study drugs
3. Known or suspected significant hypersensitivity, intolerance, or allergy to rezatapopt, metformin, rosuvastatin, repaglinide, or midazolam or any of their excipients or medicinal products with similar chemical structures, food, or other substances
4. Previously untreated brain metastases, leptomeningeal metastases, or spinal cord compression due to disease. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 4 weeks prior to starting study drugs, there is no evidence of central nervous system disease progression or mild neurologic symptoms, and there is no requirement for chronic corticosteroid therapy.
5. Stroke or transient ischemic attack within 6 months before screening
6. Clinically significant, uncontrolled heart diseases currently or within the last 6 months including:

   * QTcF >470 msec obtained as the mean from 3 consecutive resting ECGs. A QTcF value corrected for wide QRS >120 msec (QTcFBBB) should be used in place of QTcF for patients with non-clinically significant wide QRS >120 msec due to a pacemaker or bundle branch block.
   * Uncontrolled hypertension
7. Active gastrointestinal disease that may interfere significantly with the absorption, distribution, metabolism, or excretion of study drug
8. History of prior organ transplant
9. Presence of other active invasive cancers other than the one treated in this study within 2 years prior to screening, except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of the uterine cervix, or other local tumors considered cured by local treatment
10. Known, active, uncontrolled hepatitis B virus infection (i.e., viral load above the limit of quantification), hepatitis C virus infection (i.e., viral load above the limit of quantification), or human immunodeficiency virus infection (viral load >400 copies/mL of blood). Patients whose viral load is controlled should be on established antiretroviral therapy for at least 4 weeks before receiving their first dose of study drugs.
11. Patients with a known KRAS single-nucleotide variation (SNV) mutation
12. Major surgery (excluding placement of vascular access) within 4 weeks of first dose of study drugs

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Metformin Cmax geometric mean ratio | Day 1 to Day 24 of Part A
  Geometric mean metformin peak concentration (Cmax) when administered with rezatapopt versus metformin alone.
Rosuvastatin Cmax geometric mean ratio | Day 1 to Day 24 of Part A
  Geometric mean rosuvastatin peak concentration (Cmax) when administered with rezatapopt versus rosuvastatin alone.
Repaglinide Cmax geometric mean ratio | Day 1 to Day 24 of Part A
  Geometric mean repaglinide peak concentration (Cmax) when administered with rezatapopt versus repaglinide alone
Midazolam Cmax geometric mean ratio | Day 1 to Day 24 of Part A
  Geometric mean midazolam peak concentration (Cmax) when administered with rezatapopt versus midazolam alone
Metformin AUC0-t geometric mean ratio | Day 1 to Day 24 of Part A
  Geometric mean metformin area under the concentration-time curve from pre-dose (time 0) to t post-dose (AUC0-t) when administered with rezatapopt versus metformin alone
Rosuvastatin AUC0-t geometric mean ratio | Day 1 to Day 24 of Part A
  Geometric mean rosuvastatin area under the concentration-time curve from pre-dose (time 0) to t post-dose (AUC0-t) when administered with rezatapopt versus rosuvastatin alone
Repaglinide AUC0-t geometric mean ratio | Day 1 to Day 24 of Part A
  Geometric mean repaglinide area under the concentration-time curve from pre-dose (time 0) to t post-dose (AUC0-t) when administered with rezatapopt versus repaglinide alone
Midazolam AUC0-t geometric mean ratio | Day 1 to Day 24 of Part A
  Geometric mean midazolam area under the concentration-time curve from pre-dose (time 0) to t post-dose (AUC0-t) when administered with rezatapopt versus midazolam alone
PK profile of metformin - area under the concentration-time curve from pre-dose (time 0) to 24 h post-dose (AUC0-24) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of metformin
PK profile of rosuvastatin - area under the concentration-time curve from pre-dose (time 0) to 24 h post-dose (AUC0-24) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rosuvastatin
PK profile of repaglinide - area under the concentration-time curve from pre-dose (time 0) to 24 h post-dose (AUC0-24) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of repaglinide
PK profile of midazolam - area under the concentration-time curve from pre-dose (time 0) to the time 24 h post-dose (AUC0-24) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of midazolam
PK profile of metformin - area under the concentration-time curve from pre-dose (time 0) to 48 h post-dose (AUC0-48) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of metformin
PK profile of rosuvastatin - area under the concentration-time curve from pre-dose (time 0) to 48 h post-dose (AUC0-48) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rosuvastatin
PK Profile of Metformin - Time of Peak Concentration (Tmax) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of metformin
PK Profile of Rosuvastatin - Time of Peak Concentration (Tmax) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rosuvastatin
PK Profile of Repaglinide - Time of Peak Concentration (Tmax) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of repaglinide
PK Profile of Midazolam - Time of Peak Concentration (Tmax) | Day 1 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of midazolam

SECONDARY OUTCOMES:
Determine the incidence and severity of adverse events to characterize the safety of rezatapopt alone or co-administered with metformin and rosuvastatin, or repaglinide and midazolam | From Day 6 to 24 of Part A
  Number of participants with adverse events, with severity assessed using CTCAE v5.0
Assess the safety and tolerability of multiple doses of rezatapopt alone or co-administered with metformin and rosuvastatin, or repaglinide and midazolam | Day 6 to 24 of Part A.
  Changes from baseline of physical examinations.
Assess the safety and tolerability of multiple doses of rezatapopt alone or co-administered with metformin and rosuvastatin, or repaglinide and midazolam | Day 6 to Day 24 of Part A
  Changes from baseline of vital signs
Assess the safety and tolerability of multiple doses of rezatapopt alone or co-administered with metformin and rosuvastatin, or repaglinide and midazolam | Day 6 to Day 24 of Part A
  Changes from baseline of clinical laboratory values
Assess the safety and tolerability of multiple doses of rezatapopt alone or co-administered with metformin and rosuvastatin, or repaglinide and midazolam | Day 6 to Day 24 of Part A
  Changes from baseline of 12 lead triplicate ECGs (electrocardiogram)
Assess the safety and tolerability of multiple doses of rezatapopt alone or co-administered with metformin and rosuvastatin, or repaglinide and midazolam | Day 6 to Day 24 of Part A
  Changes in baseline of Eastern Cooperative Oncology Group Performance Status (ECoG) using a scale of 0-5
PK profile of rezatapopt and its metabolites, M13 and M14 - peak concentration (Cmax) | Day 6 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt and its metabolites, M13 and M14.
PK profile of rezatapopt and its metabolites, M13 and M14 - area under the concentration-time curve from pre-dose (time 0) to the time t post-dose (AUC0-t) | Day 6 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt and its metabolites, M13 and M14.
PK profile of rezatapopt and its metabolites, M13 and M14 - time of peak concentration (Tmax) | Day 6 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt and its metabolites, M13 and M14.
PK profile of rezatapopt and its metabolites, M13 and M14 - area under the concentration-time curve from pre-dose (time 0) to the time 24 h post-dose (AUC0-24) | Day 6 to Day 24 of Part A
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of rezatapopt and its metabolites, M13 and M14.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Subbiah, MD, Study Chair — SCRI
Locations (5):
- United States (5):
  - HealthOne Denver, Denver, Colorado
  - Florida Cancer Specialists, Orlando, Florida
  - SCRI Oncology Partners, Nashville, Tennessee
  - SCRI at Mary Crowley, Dallas, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No